CLINICAL TRIAL: NCT04320277
Title: Baricitinib Combined With Antiviral Therapy in Symptomatic Patients Infected by COVID-19: an Open-label, Pilot Study
Brief Title: Baricitinib in Symptomatic Patients Infected by COVID-19: an Open-label, Pilot Study.
Acronym: BARI-COVID
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital of Prato (Other)
Responsible Party: Principal Investigator, Fabrizio Cantini, Head of Rheumatology Department, Principal investigator, Hospital of Prato
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HPrato-3
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pharmacological Action
Keywords: COVID-19; Baricitinib; Moderate disease; Infection
MeSH Terms: conditions — COVID-19; Infections | interventions — baricitinib; Lopinavir; Ritonavir; BID protein, human

STUDY DESIGN:
Intervention Model Description: Patients. All consecutive patients with mild to moderate COVID-19 infection, older than 18, Patients should present fever, cough and myalgia and weakness and radiological findings of pneumonia.
  Controls. All consecutive patients with mild to moderate COVID-19 infection, older than 18, admitted during the previous 2 weeks, who were treated with antiviral and/or hydroxychloroquine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): All patients received baricitinib combined to antiviral therapy lopinavir/ritonavir for 2 weeks.
  Interventions: Drug: Baricitinib
- Controls (Active Comparator): All consecutive patients with mild to moderate COVID-19 infection, older than 18, a during the previous 2 weeks, who were treated with antiviral and/or hydroxychloroquine.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Baricitinib 4 mg/day/orally combined to antiviral therapy ritonavir for 2 weeks. Baricitinib tablets 4 mg were administered in the morning.
  Other Names: Lopinavir/Ritonavir tablets 250 mg/bid

SUMMARY:
There is no specific antiviral treatment recommended for COVID-19, and no vaccine is currently available. Baricitinib, an anti-Janus kinase inhibitor (anti-JAK) acting against JAK1 and JAK2. The drug was found capable to reduce or interrupt the passage of the virus into target cells, and to inhibit the JAK1- and JAK2-mediated cytokine release. The drug was licensed for the treatment of rheumatoid arthritis at the daily dose of 4 mg/orally, with excellent results in terms of clinical response and a good safety profile. Since baricitinib does not interact with antivirals due to its prevalent renal elimination, it may be used in combination.The evidence on the advantageous action of baricitinib on viral entry and cytokine outbreak constituted the rationale to perform a trial on patients with mild to moderate COVID-19 infection receiving baricitinib combined with antiviral therapy.

DETAILED DESCRIPTION:
Study design. Interventional, open-label, 2-week, prospective trial of a cohort of patients with mild to moderate COVID-19 infection.

Objectives. Primary. To assess the efficacy of baricitinib combined with antiviral therapy in patients with COVID-19-related mild and moderate disease in terms of reduction of the percentage of subjects requiring ICU admission.

Secondary objectives. To describe the clinical findings in a cohort of symptomatic COVID-19-infected subjects; to investigate the role of CRP, IL-6, and TNFα levels as predictor of progression to ARDS; to assess the type and incidence of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with mild to moderate COVID-19 infection
* Age >18 years,
* Clinical diagnosis of COVID19 infection
* Patients should present fever, cough and myalgia and weakness and radiological findings of pneumonia.
* All patients should be willing and able to provide written informed consent prior to performing study procedures.

Exclusion Criteria:

* Age less than 18
* History of thrombophlebitis.
* Patient with latent tuberculosis infection (Quantiferon test).
* Pregnancy and lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-16 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients requiring transfer to ICU as compared with the rate of transfers observed in controls. | 2 weeks
  The percentage of ICU admission in patients and controls will be compared for statistical difference

SECONDARY OUTCOMES:
The percentage of patients achieving the remission; CRP, IL-6 and TNFα values at baseline and during the treatment course; the number of AEs. | 2 weeks
  CRP values will be evaluated for prediction of disease worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Cantini, MD, Study Director — Hospital of Prato, Italy
Locations (1):
- Fabrizio Cantini, Prato, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Richardson P, Griffin I, Tucker C, Smith D, Oechsle O, Phelan A, Rawling M, Savory E, Stebbing J. Baricitinib as potential treatment for 2019-nCoV acute respiratory disease. Lancet. 2020 Feb 15;395(10223):e30-e31. doi: 10.1016/S0140-6736(20)30304-4. Epub 2020 Feb 4. No abstract available. PMID 32032529
- [Background] Bechman K, Subesinghe S, Norton S, Atzeni F, Galli M, Cope AP, Winthrop KL, Galloway JB. A systematic review and meta-analysis of infection risk with small molecule JAK inhibitors in rheumatoid arthritis. Rheumatology (Oxford). 2019 Oct 1;58(10):1755-1766. doi: 10.1093/rheumatology/kez087. PMID 30982883
- [Background] Stebbing J, Phelan A, Griffin I, Tucker C, Oechsle O, Smith D, Richardson P. COVID-19: combining antiviral and anti-inflammatory treatments. Lancet Infect Dis. 2020 Apr;20(4):400-402. doi: 10.1016/S1473-3099(20)30132-8. Epub 2020 Feb 27. No abstract available. PMID 32113509
- [Derived] Benucci M, Damiani A, Infantino M, Manfredi M, Quartuccio L. Old and new antirheumatic drugs for the treatment of COVID-19. Joint Bone Spine. 2020 May;87(3):195-197. doi: 10.1016/j.jbspin.2020.03.013. No abstract available. PMID 32321635